CLINICAL TRIAL: NCT05591521
Title: Evaluation of Pain in the Course of in Vitro Fertilization: the Endalgofiv-2 Study
Acronym: ENDALGOFIV-2
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2022_0015; 2022-A01468-35 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2022-08-11; First posted 2022-10-24 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Infertility
Keywords: Infertility; In Vitro Fertilization; Endometriosis; pain evaluation
MeSH Terms: conditions — Infertility; Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Using different survey to evaluate pain — Survey will be at different time of the IVF protocol (at the first medical appointment in the medically assisted department, after stimulation, after oocytes retrieval, after embryo transfer, one month after the IVF protocol)

SUMMARY:
The ENDALGOFIV study of pain assessment during the IVF pathway at Lille University Hospital, conducted from November 2018 to July 2020, showed that endometriosis patients have intense pain, particularly of a neuropathic nature, even before starting their IVF pathway compared to patients without endometriosis, but without an increase in pain scores during the IVF pathway. As a result of this study, a new pain management protocol for all patients undergoing IVF have been implemented in our MPA center. The study will be evaluated the impact of this new management.

Main objective To evaluate the effect of the change in pain management protocol in all patients (endometriotic or not) undergoing IVF treatment during the study period by comparing them to the data of the ENDALGOFIV 1 study.

ELIGIBILITY:
Inclusion Criteria:

* All patients who start an IVF cycle in the medically assisted procreation department of the Jeanne de Flandres Hospital (CHRU Lille)

Exclusion Criteria:

* Previously enrolled patient (ENDALGOFIV or ENDALGOFIV 2)
* Refusal to participate in the study
* Minor patient
* Patient over 43 years old
* BMI patient > 35
* Pregnant woman
* Unable to provide clear information to the patient
* Patient under guardianship or lack of health cover
* Patient in IVF with donation of oocyte
* IVF patients for oocyte preservation
* Patient who had already participated in the study

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — All patients who start an IVF cycle in the medically assisted procreation department of the Jeanne de Flandres Hospital (CHRU Lille)
Study Population: All patients who start an IVF cycle in the medically assisted procreation department of the Jeanne de Flandre Hospital (CHRU Lille)
Sampling Method: Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2022-11-30 (Actual); Primary Completion 2024-03-24 (Actual); Study Completion 2024-03-24 (Actual)

PRIMARY OUTCOMES:
Questionnaire douleur Saint Antoine (QDSA) | After puncture, before discharge from hospital (assessed up to 24 hours)
  QDSA for emotional and sensory dimension of pain. It's a word list to describe a pain, patient must specify the type of pain that she usually feels for 8 days by putting a cross for the correct answer (0 to 4: absent, weak, moderate, strong, extremely strong). Scored from 0 to 64

SECONDARY OUTCOMES:
Questionnaire douleur Saint Antoine (QDSA) | At baseline and during procedure ( an average up to 6 weeks)
  compare the evolution of pain during study between the 2 groups endometriosis - non endometriosis
EN = numerical scale of pain | At baseline and during procedure ( an average up to 6 weeks)
  from 0 to 10 (0 is "no pain" and 10 is "maximum pain imaginable") compare the evolution of pain during study between the 2 groups endometriosis - non endometriosis
DN4 | At baseline and during procedure ( an average up to 6 weeks)
  emotional and sensory dimension of pain, neuropathic pain survey in four questions - score on 7 compare the evolution of pain during study between the 2 groups endometriosis - non endometriosis
HAD,anxiety and depression | At baseline and during procedure ( an average up to 6 weeks)
  2 scores on 21 - "circle the number that best fits your condition" Compare the evolution of pain during study according to the 2 periods (ENDALGOFIV 1 patients and patients who benefited from the new management protocol)
EQ-5D quality of life | At baseline and during procedure ( an average up to 6 weeks)
  overall score on a numeric scale "check the box that best describes your health today", 5 themes (mobility, autonomy of the person, common activities, pain / discomfort, anxiety / depression) Compare the evolution of pain during study according to the 2 periods (ENDALGOFIV 1 patients and patients who benefited from the new management protocol)
pain catastrophism scale (PCS) | At baseline and during procedure ( an average up to 6 weeks)
  score between 0 to 52. Compare the evolution of pain during study according to the 2 periods (ENDALGOFIV 1 patients and patients who benefited from the new management protocol)
willingness to go the pain consultation: yes or no answer | during the stimulation period (an average 10 days)
  measure the impact of the pain on the pregnancy project and on the analgesic management after stimulation between the 2 endometriosis - non-endometriosis groups
willingness to take a antalgic medication during the stimulation: yes or no answer | during the stimulation period (an average 10 days)
  measure the impact of the pain on the pregnancy project and on the analgesic management after stimulation between the 2 endometriosis - non-endometriosis groups
willingness to take a antalgic medication during the punction: yes or no answer | during the stimulation period (an average 10 days)
  measure the impact of the pain on the pregnancy project and on the analgesic management after stimulation between the 2 endometriosis - non-endometriosis groups

CONTACTS AND LOCATIONS:
Overall Officials: Chrystele Rubod, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Jeanne de Flandre Chu Lille, Lille, France